CLINICAL TRIAL: NCT02815358
Title: Effects of Segmental Stabilization on the Anticipatory Postural Adjustment of Subjects With Lumbar Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 923.642
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Lumbar Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Segmental Stabilization Group (Experimental): Patients receiving segmental stabilization exercises.
  Interventions: Other: Segmental Stabilization Exercises
- Control Group (Active Comparator): Patients receiving home exercises.
  Interventions: Other: Home Exercises

INTERVENTIONS:
Other: Segmental Stabilization Exercises — The stabilization program focuses on the reestablishment of motor control and coordination between deep and superficial trunk muscles. The exercise program is based on the following criteria progression: 1) Precise contraction of the transverse abdominal and multifidus muscles, keeping the lumbar spine in a neutral position (as the middle way between maximum flexion and extension, repeated three times); 2) Keep the neutral position for 10 repetitions of 10 seconds; 3) Perform exercises with lower limbs in different postures.
  Arms: Segmental Stabilization Group
Other: Home Exercises — Home exercises include passive stretching and active mobilization of the spine.
  Arms: Control Group

SUMMARY:
This study aims to verify the effects of a segmental stabilization exercise program on the anticipatory postural adjustment of subjects with chronic lumbar pain. The effects will be assessed by means of superficial electromyography focused on the registry of the onset of multifidius and deltoid (anterior and posterior) activity during a repetitive shoulder ﬂexion/extension.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 18 and 65 years old
* chronic lumbar pain (at least 3 months)
* average pain intensity of ≥3 on a 10-point scale

Exclusion Criteria:

* presence of red flags (i.e.,tumor, known fractures, diagnosed inflammatory joint disease, etc);
* history of back surgery
* pregnancy
* less than 3 months of therapeutic treatment (physiotherapy) for low back pain

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Anticipatory Postural Adjustment by means of Electromyography | change from pre to post-treatment (8 weeks)
  Assessed by means of superficial electromyography

SECONDARY OUTCOMES:
Disability level via the Oswestry Low Back Pain Questionnaire | change from pre to post-treatment (8 weeks)
Fear of pain and avoidance of physical activity via the Fear-avoidance beliefs Questionnaire | change from pre to post-treatment (8 weeks)
Prognosis or risk of poor clinical outcome via the STarT Back Screening Tool | change from pre to post-treatment (8 weeks)
Pain level via visual analogue scale | change from pre to post-treatment (8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil